CLINICAL TRIAL: NCT03830853
Title: The Impact of Coronary Chronic Total Occlusion Percutaneous Coronary Intervention on Culprit Vessel Physiology
Acronym: IMPACT-CTO-2
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 240138
Record Dates: First submitted 2019-01-22; First posted 2019-02-05 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: CTO - chronic total occlusion; OCT - optical coherence tomography; coronary physiology; absolute flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Successful CTO PCI achieved: Patients will have successful CTO PCI (chronic total occlusion percutaneous coronary intervention) followed by physiological and intracoronary imaging. These measurements will be repeated at a 3 month follow up angiogram procedure.

SUMMARY:
Following successful CTO PCI, a multitude of physiological and anatomical changes take place. Contemporary techniques such as dissection/re-entry or lumen-lumen wiring may influence the immediate and longer term follow up of these features. It is not known whether changes in this level of physiology and anatomy in the context of CTO vessels correlate with each other, or with quality of life and exercise capacity.

This study aims to take physiological measurements of absolute coronary flow, resistance and pressure and intra-coronary imaging immediately after successful CTO PCI. The investigators will relate these to each other and to the method of revascularisation, comparing changes in these groups at three months follow up.

QoL measurements, and exercise testing will be carried out to see if there is a relationship between physiological and anatomical changes with exercise capacity and quality of life.

Results from this study could shed light on optimisation of CTO PCI procedural and clinical outcomes.

DETAILED DESCRIPTION:
Following successful chronic total occlusion (CTO) percutaneous coronary intervention (PCI), a multitude of physiological and anatomical changes take place. Contemporary techniques such as dissection/re-entry or lumen-lumen wiring may influence the immediate and longer term follow up of these features. It is not known whether changes in this level of physiology and anatomy in the context of CTO vessels correlate with each other, or with quality of life and exercise capacity.

This study aims to take physiological measurements of absolute coronary flow, resistance and pressure and intra-coronary imaging immediately after successful CTO PCI. The investigators will relate these to each other and to the method of revascularisation, comparing changes in these groups at three months follow up.

Quality of life measurements, and exercise testing will be carried out to see if there is a relationship between physiological and anatomical changes with exercise capacity and quality of life.

Results from this study could shed light on optimisation of CTO PCI procedural and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Presence of a coronary chronic total occlusion (CTO) scheduled for elective percutaneous coronary angioplasty (PCI)
* Evidence of viability in the CTO Territory

Exclusion Criteria:

* < 18 year of age
* Unable to give informed consent
* Known severe chronic kidney disease (creatinine clearance ≤30 mL/min), unless the patient is on dialysis
* Unable to receive antiplatelets or periprocedural anticoagulation
* Contraindications to adenosine
* Any study lesion characteristic resulting in the expected inability to deliver FD-OCT catheter at the distal vessel post CTO PCI (e.g. moderate or severe vessel calcification or tortuosity)
* Pregnancy, planning pregnancy during study period, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been selected for elective percutaneous coronary angioplasty (PCI) of their chronic total occlusion (CTO) as part of routine standard of care will be approached for the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change in coronary flow | 3 months
  change in coronary flow at baseline and follow up
Change in coronary resistance | 3 months
  change in coronary absolute resistance at baseline and follow up

SECONDARY OUTCOMES:
Change in coronary anatomy | 3 months
  To identify intracoronary anatomical features between baseline and follow up.
Change in exercise work load | 3 months
  Change in exercise work measured in METS (metabolic equivalents).
Change in quality of life | 3 months
  change in quality measured by the validated Seattle angina seven question questionnaire from baseline to follow up. This is a scale based on 7 questions giving scores of 0-100 on physical limitation, angina, and quality of life, with the average of these scores giving a mean value also ranging from 0-100 of the overall summary score.
Change in coronary pressure measurements | 3 months
  change in fractional flow reserve (FFR) at baseline and follow up

CONTACTS AND LOCATIONS:
Overall Officials: John Davies, MBBS, PhD, Principal Investigator — Basildon and Thurrock University Hospitals
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No